CLINICAL TRIAL: NCT03982407
Title: Pilot Study of Integrated Time-of-Flight (TOF) 68 GA-PSMA - Gadoxetate PET/MR for Evaluation of Hepatocellular Carcinoma
Brief Title: 68 Ga PSMA PET/MRI for Hepatocellular Carcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ajit H. Goenka, MD (Other)
Responsible Party: Sponsor-Investigator, Ajit H. Goenka, MD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-011263; NCI-2019-08426 (Other: NCI); MC1944 (Other: Mayo Clinic)
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga68 PSMA PET-MR (Experimental): 68Ga labeled PSMA -11 (or PSMA-HBED_CC) PET/MRI scan
  Interventions: Drug: 68Ga-PSMA-11 PET/MRI

INTERVENTIONS:
Drug: 68Ga-PSMA-11 PET/MRI — The PET/MRI exam-related patient visit will last approximately 2 to 2.5 hours, including 30-minute nursing assessment, 45-60 minutes for PSMA uptake and 60 minutes for PET/MRI scan. They will be contacted within the next 72 hours to complete a brief phone survey.

SUMMARY:
This is a pilot study to investigate the evaluate to use of a drug/radiopharmaceutical called Gallium-68 PSMA-11 (68Ga-PSMA-11) for use in PET/MRI evaluation of hepatocellular carcinoma

DETAILED DESCRIPTION:
This is a prospective pilot proof-of-concept single-center study. Primary Objective Using surgical histopathology as the reference standard, the investigators intend to achieve the following objectives in adult subjects with Hepatocellular Carcinoma (HCC) undergoing surgical resection or transplant:

1. To demonstrate the feasibility of 68Ga-PSMA-PET/MRI for imaging patients with HCC
2. To estimate the sensitivity of SUVmax on PSMA PET for identification of LI-RADS® 5 (definitely HCC) observations or biopsy proven HCC(s).
3. To perform a Radiology-Pathology correlation of PSMA uptake at PET with HCC tumor PSMA immunostaining, tumor pathology features, and signal and enhancement characteristics at MRI

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk for HCC with either an imaging diagnosis of HCC by ceCT or ceMRI (LI-RADS 5) confirmed by a board-certified abdominal radiologist or biopsy-proven HCC confirmed by a hepatobiliary pathologist
* No prior treatment for HCC
* Subjects who are expected to undergo surgical resection of the hepatic lesion(s) and/or liver transplant
* Male or female with age greater than 18 years, with the capacity to give informed consent and willingness to provide a written consent.

Exclusion Criteria:

* Subjects requiring emergent surgery for a ruptured/bleeding HCC
* Bilirubin > 3.0 mg/dL, which is a contraindication for Gadoxetate, the MRI contrast agent
* Pregnant and/or breast-feeding subjects. A negative pregnancy test within 48 hours of the PET scan.
* Subjects with higher than the weight/size limitations of PET/MRI scanner.
* Subjects with contraindication to MRI including: Subjects who have a heart pacemaker, subjects who have a metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain, subjects who have implanted devices with magnets, subjects who have other implanted electronic devices, subjects who have deep brain stimulator, subjects who have vagal nerve stimulator, subjects with cochlear (ear) or auditory implants
* Subjects with history of allergic response to radiocontrast media
* Subjects with known history of claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of PSMA PET-MR for identification of intra and extrahepatic hepatocellular carcinoma in patients | 18 months
  Sensitivity of PSMA PET-MRI for detection of LI-RADS 5 (definitely HCC) lesions on a per-lesion basis with histopathology as the gold standard. We will perform a Radiologic-pathologic correlation comparing HCC PSMA SUVmax with tumor PSMA immunostaining positivity.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit H Goenka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials